CLINICAL TRIAL: NCT02073565
Title: Japan-USA Harmonized Assessment by Randomized, Multi-Center Study of OrbusNEich's Combo StEnt (Japan-USA HARMONEE): Assessment of a Novel DES Platform For Percutaneous Coronary Revascularization in Patients With Ischemic Coronary Disease and NSTEMI Acute Coronary Syndrome
Brief Title: HARMONEE - Japan-USA Harmonized Assessment by Randomized, Multi-Center Study of OrbusNEich's Combo StEnt
Acronym: HARMONEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OrbusNeich (Industry)
Collaborators: OrbusNeich Medical K.K. (Unknown); Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VP-0601; OMKK 02 (Other: Japan PMDA)
Record Dates: First submitted 2014-02-13; First posted 2014-02-27 (Estimated); Results first posted 2018-11-21 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-04

CONDITIONS: Coronary Arteriosclerosis; Non ST Segment Elevation Acute Coronary Syndrome
Keywords: intracoronary stent; drug eluting stent; sirolimus; endothelial progenitor cells
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combo (Experimental): The Combo Stent is composed of the OrbusNeich R stent™, with an abluminal coating of a bioabsorbable polymer matrix formulated with sirolimus for sustained release, and an anti-CD34 antibody cell capture coating on the luminal surface.
  Interventions: Device: OrbusNeich Combo stent™
- Everolimus Eluting Stent (EES) (Active Comparator): Everolimus Eluting Stent (EES) (Xience V, Xience Prime, Xience Xpedition stents, Abbott Vascular/Abbott Vascular Japan). Xience Prime inherited the clinical result of Xience V and is a product that obtains efficiency essentially equal to Xience V.
  Interventions: Device: Everolimus Eluting Stent (EES)

INTERVENTIONS:
Device: OrbusNeich Combo stent™ — The Combo Stent is composed of the OrbusNeich R stent™, with an abluminal coating of a bioabsorbable polymer matrix formulated with sirolimus for sustained release, and an anti-CD34 antibody cell capture coating on the luminal surface.
  Arms: Combo
Device: Everolimus Eluting Stent (EES) — Everolimus Eluting Stent (EES) (Xience V, Xience Prime, Xience Xpedition stents, Abbott Vascular/Abbott Vascular Japan). Xience Prime inherited the clinical result of Xience V and is a product that obtains efficiency essentially equal to Xience V.
  Arms: Everolimus Eluting Stent (EES)

SUMMARY:
This is a multi-center, single-blind, randomized, active-controlled, clinical trial in Percutaneous Coronary Intervention (PCI) subjects. Subjects will be randomized to receive the Combo stent as the investigational treatment arm or an Everolimus Eluting Stent (EES) as the active-control arm.

DETAILED DESCRIPTION:
Up to 50 sites are proposed in Japan and the United States to enroll 286 subjects (271 evaluable) in each of 2 arms, for a total sample size of 572 subjects (542 evaluable) who are admitted to the hospital for a planned (elective and urgent) percutaneous coronary artery intervention procedure.

After stent implantation, subjects will be contacted for follow-up at 30 days; 6 months; and 1, 2, 3, 4, and 5 years. At 12 months a clinical evaluation will be completed before cardiac catheterization and angiographic assessment.

Rationale: This study is intended to demonstrate that the Combo stent platform shows superiority to an imputed Bare Metal Stent (BMS) performance goal, noninferior effectiveness and safety vs best-in-class second-generation everolimus-eluting stent (EES) (Xience V, Xience Prime, Xience Xpedition stents; [Abbott Vascular/Abbott Vascular Japan]), and evidence of mechanistic activity of the anti-CD34-Ab endothelial progenitor cell (EPC) capture technology with healthy level of intimal tissue coverage superior to that of the best-in-class EES.

To ensure the robustness and interpretability of results, the current proposal includes a number of unique design features:

* Largest randomized Drug-Eluting Stent (DES) study ever performed in Japan
* Enriched population, including stabilized Non-ST-elevation myocardial infarction (NSTEMI) subjects with greater likelihood of plaque rupture associated with their clinical syndromes
* Collaboration between with Japan and the United States as a "Proof of Concept" program under the auspices of the Harmonization by Doing Initiative, Working Group 1 (WG 1), including concomitant enrollment in U.S.A. sites as an FDA-approved Investigational Device Exemption (IDE) study
* Head-to-head randomization against state-of-the-art EES platform control, analyzed for clinical noninferiority
* Statistical analysis vs imputed BMS analyzed for clinical superiority
* Fractional flow reserve (FFR) follow-up of 100% of subjects enrolled, providing clinically relevant physiologic assessment of all subjects for 1 year ischemia-driven Target Vessel Revascularization (TVR) analysis
* Mechanistic Optical coherence tomography (OCT) imaging observations in 140 subjects using 6 French catheters as follows:

  * Cohort A (30 subjects, 1:1 Combo and EES): Mechanistic imaging observations to provide serial 6 month and 1 year OCT evaluation of healthy intimal tissue coverage, intracoronary thrombosis, and stent malapposition and quantitative coronary angiographic (QCA) analysis to assess 1 year late loss.
  * Cohort B (110 subjects, 1:1 Combo and EES): Mechanistic imaging observations to assess 1 year OCT evaluation of healthy intimal tissue coverage, intracoronary thrombosis, and stent malapposition, and QCA analysis to assess 1 year late loss. Combined with the 12 month imaging of Cohort A, this study will provide OCT and QCA observations at 1 year in 140 patients, half with Combo and half with EES.
  * Cohort C: 432 subjects (216 subjects per arm) will undergo all clinical follow-up assessments with FFR and angiographic assessments at 12 months. Cohort C will be the last cohort to enroll.
* In the 110 subjects in Cohort B, 30 day and 1 year human antimurine antibody (HAMA) titers will also be collected.

ELIGIBILITY:
Inclusion Criteria

To be eligible for this trial, subjects must meet all of the following criteria:

1. Subject is able to verbally confirm understanding of risks, benefits, and treatment alternatives of Combo vs EES stent, and the subject or a legally authorized representative (LAR) must provide written informed consent before any study-related procedures are performed.
2. Subject must be at least 20 years of age at the time of randomization.
3. Subject must have clinical or functional evidence of myocardial ischemia (eg, stable or unstable angina, stabilized non-ST-elevation myocardial infarction confirmed by serum markers, ischemia by positive functional study, abnormal FFR, or a reversible change in the electrocardiogram (ECG) consistent with ischemia).
4. Subject must be acceptable candidate with anatomy suitable for PCI with a DES.
5. Subject agrees to return for all study-related follow-up assessments, including invasive OCT follow-up assessment at 6 months (Cohort A) and at 1 year postprocedure (Cohorts A, B, and C).
6. Subject is an acceptable candidate for Coronary artery bypass grafting (CABG) surgery.

   Angiographic Anatomy Criteria-
7. Target lesions must be located in a native coronary artery with visually estimated diameter of 2.5 mm to 3.5 mm, inclusive, and up to 3 de novo target lesions may be treated, with a maximum of 2 de novo target lesions per epicardial vessel, with a maximum of 2 target vessels.
8. Target lesions should be treatable with a single stent, and must measure 28 mm or less in length by visual estimation (2 mm or more of nondiseased tissue on either side of the target lesion should be covered by the study stent).
9. If more than 1 target lesion will be treated, the reference vessel diameter and lesion length of each target lesion must meet the above criteria.
10. Target lesions must be in a major artery or branch with a visually estimated stenosis of 50% or greater and less than 100% with a Thrombolysis in Myocardial Infarction (TIMI) flow of 1 or greater.
11. Previous percutaneous intervention of lesions in a target vessel (including side branches) is allowed if done 9 or more months before the study procedure and greater than 10 mm from the current target lesion.
12. Nonstudy percutaneous interventions for lesions in a nontarget vessel are allowed if done 9 or more months before the study procedure, in the absence of documented ischemia or angiographic restenosis related to the vessel.

Exclusion Criteria

If a subject meets any of the following criteria, he or she may not be enrolled in the study:

1. ST-Elevation Myocardial Infarction (STEMI) at index presentation or within 7 days of study screening.
2. Subject has current unstable arrhythmias or intractable angina with ECG changes or shock requiring pressors or mechanical assist device (intraaortic balloon pump, left ventricular assist device, Impella, etc.).
3. Subject has known left ventricular ejection fraction (LVEF) less than 30%.
4. Subject has received a heart transplant or any other organ transplant or is on a waiting list for any organ transplant.
5. Subject is receiving or scheduled to receive anticancer therapy for malignancy within 30 days before or after the procedure.
6. Subject is receiving immunosuppression therapy, has known serious immunosuppressive disease (eg, human immunodeficiency virus), or has severe autoimmune disease that requires chronic immunosuppressive therapy (eg, systemic lupus erythematosus).
7. Subject has known hypersensitivity or contraindication to aspirin; both heparin and bivalirudin; all available P2Y12 inhibitors (clopidogrel, prasugrel, ticlopidine, and ticagrelor); any everolimus, sirolimus, cobalt, chromium, nickel, tungsten, acrylic, or fluoro polymers; or hypersensitivity to contrast media that cannot be adequately premedicated.
8. Subject has previously received murine therapeutic antibodies and exhibited sensitization through the production of human anti-mouse antibodies (HAMAs).
9. Subject has elective surgery planned within the first 12 months after the procedure that will require interruption or discontinuation of planned Dual Antiplatelet Therapy (DAPT).
10. Subject has known platelet count less than 100,000 cells/mm3 or greater than 700,000 cells/mm3, a white blood cell count of less than 3000 cells/mm3, or documented or suspected liver disease (including laboratory evidence of hepatitis).
11. Subject has known renal insufficiency (eg, serum creatinine level of greater than 2.5 mg/dL or subject is on dialysis).
12. Subject has history of bleeding diathesis or coagulopathy or will refuse blood transfusions.
13. Subject has had a cerebrovascular accident or transient ischemic neurological attack within the past 6 months.
14. Subject has had a significant gastrointestinal or urinary bleed within the past 6 months.
15. Subject has known extensive peripheral vascular disease that precludes safe 6 French sheath insertion.
16. Known other medical illness (eg, cancer, chronic infectious disease, severe vascular disease, or congestive heart failure) or known history of substance abuse (alcohol, cocaine, heroin, etc.) that may cause noncompliance with the protocol, confound the data interpretation, or is associated with a life expectancy of less than 1 year.
17. Currently participating in another clinical study that has not yet reached its primary endpoint.
18. Currently pregnant or breast-feeding or is planning pregnancy in the period up to 1 year following index procedure. Female subjects of childbearing potential must have a negative pregnancy test within 7 days before the index procedure.

    Angiographic Exclusion Criteria-

    If the target lesion meets any of the following criteria, the subject may not be enrolled in the study:
19. Unprotected left main coronary artery location.
20. Unprotected ostial (located within 2 mm of the origin) left anterior descending artery or left circumflex.
21. Located within an arterial or saphenous vein graft or graft anastomosis, distal to a diseased arterial or saphenous vein graft (visually estimated graft diameter stenosis greater than 40%).
22. Involves a bifurcation in which the side branch is 2 mm or greater in diameter AND would be covered by the planned stent.
23. Involves a side branch requiring predilation.
24. Total occlusion (TIMI flow 0) before wire crossing.
25. Extreme tortuosity proximal to or within the lesion.
26. Extreme angulation (90º or greater) proximal to or within the lesion.
27. Heavy calcification, defined as multiple persisting opacifications of the coronary wall visible in more than one projection surrounding the complete lumen of the coronary artery at the site of the lesion.
28. Restenotic vessel from previous intervention.
29. Received brachytherapy in any epicardial vessel (including side branches).
30. Target vessel contains angiographically visible thrombus.
31. Serial lesions or diffuse disease with high probability of bailout requiring 3 or more stents in a single vessel, more than 5 stents per subject, or more than 2 vessels.
32. Target or nontarget vessel lesion (including all side branches) is present with a high probability of requiring PCI within 12 months after the index procedure.
33. Stent overlapping is a planned treatment of the target lesion.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 572 (Actual)
Dates: Start 2014-02; Primary Completion 2017-07-14 (Actual); Study Completion 2021-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell W Krucoff, MD, Principal Investigator — Duke Clinical Research Institute; Shigeru Saito, MD, Principal Investigator — Shonan Kamakura General Hospital
Locations (50):
- United States (17):
  - MedStar Clinical Research Center, Washington D.C., District of Columbia
  - Atlantic Clinical Research Collaborative-Cardiology, Lake Worth, Florida
  - University of Miami, Miami, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - North Georgia Heart Foundation, Gainesville, Georgia
  - Maine Medical Center, Portland, Maine
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Lahey Clinic, Burlington, Massachusetts
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Mount Sinai Medical Center, New York, New York
  - University of Rochester Medical Center-Strong Memorial Hospital, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - The Ohio State University Medical Center, Columbus, Ohio
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Japan (33):
  - Saiseikai Fukuoka General Hospital, Fukoka-shi, Fukuoka
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Shinkoga Hospital, Kurume-shi, Fukuoka
  - Tsuchiya General Hospital, Hiroshima, Hiroshima
  - Hakodate Municipal Hospital, Hakodate-shi, Hokkaido
  - Sapporo Higashi Tokushukai Hospital, Sapporo, Hokkaido
  - Hyogo Brain and Heart Centre, Himeji-shi, Hyōgo
  - Takahashi Hospital, Kobe, Hyōgo
  - Higashi Takarazuka Satoh Hospital, Takarazukasi, Hyōgo
  - Tsuchiura Kyodo Hospital, Tsuchiura, Ibaraki
  - Kanazawa Cardiovascular Hospital, Kanazawa, Ishikawa-ken
  - National Hospital Organisation Kagoshima Medical Centre, Kagoshima, Kagoshima-ken
  - Shonan Kamakura General Hospital, Okamoto, Kamakura City
  - Kanto Rosai Hospital, Kawasaki-shi, Kanagawa
  - Saiseikai Yokohamashi Tobu Hospital, Yokohama, Kanagawa
  - Kyoto-Katsura Hospital, Kyoto, Kyoto
  - Miyazaki Medical Association Hospital, Miyazaki, Miyazaki
  - Kurashiki Central Hospital, Kurashiki-shi, Okayama-ken
  - The Sakakibara Heart Institute of Okayama, Okayama, Okayama-ken
  - Sakurabashi Watanabe Hospital, Osaka, Osaka
  - Osaka Saiseikai Nakatsu Hospital, Osaka, Osaka
  - Saga University Hospital, Saga, Saga-ken
  - Saitama Prefectural Cardiovascular and Respiratory Disease Centre, Kumagaya-shi, Saitama
  - Okamura Memorial Hospital, Suntou-gun, Shizouka
  - Jichi Medical University Hospital, Shimotsuke-shi, Tochigi
  - Department of Cardiovascular Medicine, Juntendo University School of Medicine, Bunkyo-ku, Tokyo
  - Sakakibara Memorial Hospital, Fuchu-shi, Tokyo
  - Teikyo University Hospital, Itabashi-ku, Tokyo
  - Toho University Ohashi Hospital, Meguro-ku, Tokyo
  - The Cardiovascular Institute Hospital, Minato-ku, Tokyo
  - Showa University Hospital, Shinagawa-ku, Tokyo
  - Cardiac Catheterisation Laboratory, Keio University School of Medicine, Shinjuku-ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo

REFERENCES:
- [Background] Kong DF, Saito S, Nakamura S, Mehran R, Rowland SM, Handler A, Al-Khalidi HR, Krucoff MW. Rationale and design of the Japan-USA harmonized assessment by randomized, multicenter study of OrbusNEich's combo StEnt (Japan-USA HARMONEE): Assessment of a novel DES platform for percutaneous coronary revascularization in patients with ischemic coronary disease and non-ST-elevation acute coronary syndrome. Am Heart J. 2017 May;187:112-121. doi: 10.1016/j.ahj.2017.02.004. Epub 2017 Feb 12. PMID 28454795
- [Result] Saito S, Krucoff MW, Nakamura S, Mehran R, Maehara A, Al-Khalidi HR, Rowland SM, Tasissa G, Morrell D, Joseph D, Okaniwa Y, Shibata Y, Bertolet BD, Rothenberg MD, Genereux P, Bezerra H, Kong DF. Japan-United States of America Harmonized Assessment by Randomized Multicentre Study of OrbusNEich's Combo StEnt (Japan-USA HARMONEE) study: primary results of the pivotal registration study of combined endothelial progenitor cell capture and drug-eluting stent in patients with ischaemic coronary disease and non-ST-elevation acute coronary syndrome. Eur Heart J. 2018 Jul 7;39(26):2460-2468. doi: 10.1093/eurheartj/ehy275. PMID 29931092

RESULTS

PARTICIPANT FLOW:
Period: Intention-To-Treat Subjects-Cohorts AB&C
Arm/Group | Combo | Everolimus Eluting Stent (EES)
Started | 287 | 285
Completed | 285 | 279
Not Completed | 2 | 6
Period: Cohort A
Arm/Group | Combo | Everolimus Eluting Stent (EES)
Started | 16 | 14
Completed | 15 | 14
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Cohort B
Arm/Group | Combo | Everolimus Eluting Stent (EES)
Started | 54 | 56
Completed | 53 | 54
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2
Period: Cohort C
Arm/Group | Combo | Everolimus Eluting Stent (EES)
Started | 217 | 215
Completed | 217 | 211
Not Completed | 0 | 4
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combo | Everolimus Eluting Stent (EES) | Total
Number analyzed (Participants) | 287 | 285 | 572
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (9.6) | 66.5 (10.4) | 67.0 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 73 | 149
  Male | 211 | 212 | 423
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian (non-Japanese)- | 1 | 1 | 2
  Race: Japanese | 219 | 219 | 438
  Race: Black or African American | 10 | 4 | 14
  Race: White/Caucasian | 57 | 59 | 116
  Race: Other | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 67 | 66 | 133
  Japan | 220 | 219 | 439
Non-ST-segment elevation myocardial infarction (Non-STEMI) Presentation [Count of Participants; unit: Participants] | 14 | 12 | 26
Multivessel Coronary Artery Disease (MV CAD) [Count of Participants; unit: Participants] | 33 | 31 | 64
Previous Myocardial Infarction (MI) [Count of Participants; unit: Participants] | 45 | 45 | 90
Previous Percutaneous Coronary Intervention (PCI) [Count of Participants; unit: Participants] | 72 | 83 | 155
Previous Coronary Artery Bypass Grafting (CABG) [Count of Participants; unit: Participants] | 4 | 5 | 9
Hypertension [Count of Participants; unit: Participants] | 218 | 220 | 438
Congestive Heart Failure [Count of Participants; unit: Participants] | 11 | 24 | 35
Diabetes [Count of Participants; unit: Participants]
  Diabetes: Insulin Dependent | 24 | 18 | 42
  Diabetes: Non-insulin Dependent | 93 | 75 | 168
  Participants without Diabetes | 170 | 192 | 362
Cigarette Smoking (current/former) [Count of Participants; unit: Participants] | 191 | 175 | 366
Chronic Renal Insufficiency [Count of Participants; unit: Participants] | 11 | 5 | 16
Hypercholesterolemia [Count of Participants; unit: Participants] | 225 | 227 | 452
Planned Dual Antiplatelet Therapy (DAPT) at 6 months [Count of Participants; unit: Participants] | 5 | 11 | 16
Planned Dual Antiplatelet Therapy (DAPT) at 1 year [Count of Participants; unit: Participants] | 247 | 243 | 490
Planned Statins at 1 year [Count of Participants; unit: Participants] | 233 | 228 | 461
Planned Beta-blockers at 1 year [Count of Participants; unit: Participants] | 103 | 100 | 203

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: The primary clinical endpoint of Target Vessel Failure (TVF), defined as cardiac death, target-vessel myocardial infarction (MI), or ischemia-driven Target Vessel Revascularization(TVR) by percutaneous or surgical methods, at 1 year.
Time Frame: 1 year follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Combo | Everolimus Eluting Stent (EES)
Number analyzed (Participants) | 287 | 285
Participants | 20 | 12

2. Secondary Outcome: Percentage of Healthy Tissue Coverage That Was Greater Than 40 Micrometers
Description: The secondary efficacy endpoint is mechanistic Optical coherence tomography (OCT) healthy level of intimal tissue coverage, determined by the OCT core laboratory at 1 year for subjects in Cohorts A and B. This reports the percentage of healthy tissue coverage that was great than 40 micrometers.
Time Frame: 1 year
Population: Cohorts A and B - Subjects with analyzable Optical coherence tomography (OCT) follow-up
Measure: Mean (95% Confidence Interval); unit: Healthy Tissue Strut Coverage (>40 µm) %
Units Other Than Participants: lesions
Arm/Group | Combo | Everolimus Eluting Stent (EES)
Number analyzed (Participants) | 65 | 63
Number analyzed (lesions) | 62 | 60
Healthy Tissue Strut Coverage (>40 µm) % | 91.27 [88.71 to 93.84] | 74.82 [70.02 to 79.62]

3. Other Pre Specified Outcome: Number of Patients With Clinically and Functionally Ischemia-Driven Target Lesion Revascularization (TLR)
Description: Clinically and functionally ischemia-driven target lesion revascularization (TLR), including use of target-vessel Fractional Flow Reserve (FFR), analyzed dichotomously using the Fractional Flow Reserve (FFR) vs. Angiography in Multivessel Evaluation (FAME) study criteria of 0.8 during a 2 minute infusion of adenosine or adenosine triphosphate.34 Abnormal FFR-driven interventions at 1 year will be included in the evaluation of ischemia-driven TLR.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Combo | Everolimus Eluting Stent (EES)
Number analyzed (Participants) | 287 | 285
Participants | 12 | 8

4. Other Pre Specified Outcome: Number of Patients Exhibiting Human Antimurine Antibody (HAMA) Reaction
Description: Serum will be assessed for HAMA development at index, 30 days, and 12 months in Cohort B subjects. Human antimurine antibody plasma assessment will be with blood draws performed during index procedure, 30 day follow-up visit, and 1 year catheterizations.
Time Frame: Day of device implantation, 30 days, 12 months
Population: Cohort B - Please note that for the "1 Year HAMA Responders" Row in the Combo arm, 52 participants were analyzed (1 participant withdrew and 1 participant died). For the "1 Year HAMA Responders" Row in the EES arm, 52 participants were analyzed (2 participants withdrew and 2 participants were not present for the 1 year visit).
Measure: Count of Participants; unit: Participants
Arm/Group | Combo | Everolimus Eluting Stent (EES)
Number analyzed (Participants) | 54 | 56
Participants
  Baseline HAMA Responders | 0 | 0
  30 day HAMA Responders | 0 | 0
  1 Year HAMA Responders: number analyzed (Participants) | 52 | 52
  1 Year HAMA Responders | 0 | 0

ADVERSE EVENTS:
Time Frame: Per the protocol, all adverse events will be collected from the point of subject enrollment through the 1-year follow-up. All adverse events listed as protocol-specific endpoints (Death, Cardiac death, MI, Target vessel MI, TLR (ischemia driven), TVR (ischemia driven), Stroke, transient ischemic attack (TIA), and Stent Thrombosis (ARC definition)) will be collected from 1-year follow to the completion of the study at the 5-year follow-up. The data reported below is at 1 year.
Arm/Group | Combo | Everolimus Eluting Stent (EES)
All-Cause Mortality (participants affected / at risk) | 2/287 | 0/285
Serious Adverse Events (participants affected / at risk) | 42/287 | 42/284
Other Adverse Events (participants affected / at risk) | 0/287 | 0/284
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combo (N=287) | Everolimus Eluting Stent (EES) (N=284)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 3 (4) | 0 (0)
Angina unstable (Cardiac disorders) | 2 (2) | 3 (3)
Arteriospasm coronary (Cardiac disorders) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disection (Cardiac disorders) | 1 (1) | 1 (1)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 3 (4) | 3 (3)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (2) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Catheter site erosion (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 4 (4) | 3 (3)
Vascular stent restenosis (General disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fractured ischium (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 2 (4) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vessel puncture site haemorrhage (General disorders) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood pressure decreased (Investigations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral artery occlusion (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary bladder rupture (Renal and urinary disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetes mellitus management (Surgical and medical procedures) | 1 (1) | 0 (0)
Air embolism (Vascular disorders) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Iliac artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-16): https://cdn.clinicaltrials.gov/large-docs/65/NCT02073565/Prot_SAP_000.pdf